CLINICAL TRIAL: NCT07344558
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1b Clinical Study of the Safety, Tolerability, and Pharmacokinetics of MNKD-201 (Nintedanib Dry Powder Inhalation) in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: A Study to Evaluate Safety, Tolerability and Pharmacokinetics of MNKD-201 in Patients With Idiopathic Pulmonary Fibrosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MKC-NI-002
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Nintedanib; dry powder inhalation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: MNKD-201 Target Dose or placebo (Experimental): Participants will receive a target dose of MNKD-201 (Nintedanib DPI) or placebo, administered via oral inhalation three times daily for 7 days
  Interventions: Drug: MNKD-201(Nintenadib DPI)
- Cohort 2: MNKD-201 High Dose or placebo (Experimental): Participants will receive a high dose of MNKD-201 (Nintedanib DPI) or placebo, administered via oral inhalation twice daily for 7 days
  Interventions: Drug: MNKD-201(Nintenadib DPI)
- Placebo (Placebo Comparator): Participants will receive matching placebo across both cohorts of the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MNKD-201(Nintenadib DPI) — MNKD-201 is a dry powder nintedanib formulation for oral inhalation.
  Arms: Cohort 1: MNKD-201 Target Dose or placebo; Cohort 2: MNKD-201 High Dose or placebo
Drug: Placebo — The placebo control in this study is an empty cartridge without any powder.
  Arms: Placebo

SUMMARY:
MKC-NI-002 is a Phase 1b, randomized, double-blind, placebo-controlled study of nintedanib inhalation powder (MNKD-201) in patients with Idiopathic Pulmonary Fibrosis (IPF). The trial consists of Multiple Ascending Doses (MAD) with the primary objective to evaluate safety, tolerability and pharmacokinetics (PK) of MNKD-201 compared to placebo in patients with IPF.

ELIGIBILITY:
Inclusion Criteria:

1. Is ≥40 to ≤75 years of age at the time of signing the informed consent form.
2. Diagnosis of IPF
3. Either treatment-naive or is currently on background pirfenidone on a stable dose for at least 3 months prior to Screening.
4. Has FVC >45% and <100% of predicted of normal, as determined by the central spirometry reader, during Screening.
5. DLCO corrected for hemoglobin [Visit 1] ≥40% of predicted of normal, within 12 months of Screening. If no historical DLCO is available prior to Screening, this is to be done during Screening and read locally.
6. Has a body weight >40 kg (>88 lbs.) at Screening.
7. For female participants of childbearing potential, agreement to use acceptable birth control
8. For male participants who can father a child and are having intercourse with females of childbearing potential, agreement to use a protocol-recommended method of contraception
9. Is capable of performing spirometry, as required by the study procedures and ATS guidelines.
10. CT chest within 2 years of Screening, consistent with an IPF diagnosis, per investigator assessment.

Exclusion Criteria:

1. Known explanation for interstitial lung disease, including but not limited to radiation, sarcoidosis, hypersensitivity pneumonitis, and bronchiolitis obliterans organizing pneumonia.
2. Diagnosis of any connective tissue disease, including but not limited to scleroderma/systemic sclerosis, polymyositis/dermatomyositis, systemic lupus erythematosus, and rheumatoid arthritis, regardless of whether or not it is presumed to be related to their pulmonary fibrosis diagnosis.
3. Major extrapulmonary physiological restriction (e.g., chest wall abnormality, large pleural effusion), as determined by the investigator.
4. Significant Cardiovascular diseases
5. Has had a recent or an ongoing systemic infection
6. Prior hospitalization for confirmed coronavirus disease 2019 (COVID-19), acute exacerbation of IPF or any lower respiratory tract infection within 3 months of Screening.
7. Has a history of asthma, with the exception of resolved childhood asthma.
8. Has known obstructive lung disease
9. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin >1.5 times the upper limit of normal (ULN) during Screening.
10. Advanced liver and kidney function.
11. Current or recent (within 30 days of Screening) use of nintedanib.
12. Use of prednisone ≥10 mg/day within 3 months prior to Screening, or other significant immunosuppression
13. Active lung cancer (primary or metastatic) or any cancer requiring chemotherapy or radiation therapy within 3 years, except appropriately treated non-melanoma skin cancer, localized non-malignant prostate cancer, or in situ carcinoma of uterine cervix.
14. Has participated in another clinical study of a new chemical entity, new device, or a prescription medicine within the 1 month before Screening
15. Current alcohol, medication, or illicit drug abuse
16. Has lost more than 400 mL blood, e.g., as a blood donor, or donor of blood products, during the 3 months prior to Screening.
17. Has received a live vaccine within the 3 months prior to the first dose of study drug.
18. Smokes (any substance including electronic cigarettes and marijuana) within 3 months prior to Screening or is an ex-cigarette smoker who gave up <1 year ago.
19. Has oxygen requirement of > 3 liters/min at rest.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
(Cohort 1) Events of Bronchospasm | Up to Day 7
  The within-treatment number and proportion of participants with events of bronchospasm (e.g., treatment emergent adverse events [TEAE] immediately after inhalation of wheezing or chest tightness)
(Cohort 2) Events of Bronchospasm | Up to Day 7
  The within-treatment number and proportion of participants with events of bronchospasm (e.g., treatment emergent adverse events [TEAE] immediately after inhalation of wheezing or chest tightness)
(Cohort 1) Changes in FEV1 (mL) from pre-dose to post-dose | Up to Day 7
  The within-treatment number and proportion of participants with changes in FEV1 from pre-dose to any time post-dose
(Cohort 2) Changes in FEV1 (mL) from pre-dose to post-dose | Up to Day 7
  The within-treatment number and proportion of participants with changes in FEV1 from pre-dose to any time post-dose
(Cohort 1) Changes in FEV1 / FVC ratio from pre-dose to post-dose | Up to Day 7
  The within-treatment number and proportion of participants with changes in FEV1/FVC ratio from pre-dose to any time post-dose
(Cohort 2) Changes in FEV1 / FVC ratio from pre-dose to post-dose | Up to Day 7
  The within-treatment number and proportion of participants with changes in FEV1/FVC ratio from pre-dose to any time post-dose
(Cohort 1) Rate of Study Drug Discontinuations | Up to Day 7
  The within-treatment number and proportion of participants with study drug dose discontinuations
(Cohort 2) Rate of Study Drug Discontinuations | Up to Day 7
  The within-treatment number and proportion of participants with study drug dose discontinuations
(Cohort 1) Rate of Study Drug Dose Reductions | Up to Day 7
  The within-treatment number and proportion of participants with study drug dose reductions
(Cohort 2) Rate of Study Drug Dose Reductions | Up to Day 7
  The within-treatment number and proportion of participants with study drug dose reductions
(Cohort 1) Rate of Treatment Emergent Adverse Events (TEAEs) | Up to Day 7
  The within-treatment number and proportion of participants with TEAEs overall and by severity, relationship to study drug, and outcome
(Cohort 2) Rate of Treatment Emergent Adverse Events (TEAEs) | Up to Day 7
  The within-treatment number and proportion of participants with TEAEs overall and by severity, relationship to study drug, and outcome
(Cohort 1) Rate of Treatment Related Adverse Events (TRAEs) | Up to Day 7
  The within-treatment number and proportion of participants with TRAEs overall and by severity and outcome
(Cohort 2) Rate of Treatment Related Adverse Events (TRAEs) | Up to Day 7
  The within-treatment number and proportion of participants with TRAEs overall and by severity and outcome
(Cohort 1) Rate of Serious Adverse Events (SAEs) | Up to Day 7
  The within-treatment number and proportion of participants with SAEs overall and by severity, relationship to study drug, and outcome
(Cohort 2) Rate of Serious Adverse Events (SAEs) | Up to Day 7
  The within-treatment number and proportion of participants with SAEs overall and by severity, relationship to study drug, and outcome

SECONDARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of MKND-201 in patients with IPF | Up to Day 7
  MTD within the tested MNKD-201 dose range

CONTACTS AND LOCATIONS:
Overall Officials: Wassim Fares, MD, MSc, FCCP, Study Director — Mannkind Corporation
Locations (5):
- United States (5):
  - VALDI, Fresno, California
  - Palmtree Clinical Research, Palm Springs, California
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Low Country Research, Charleston, South Carolina
  - Metroplex Pulmomary & Sleep Center, McKinney, Texas

IPD SHARING:
Plan to Share IPD: Undecided
under assessment